CLINICAL TRIAL: NCT02224573
Title: An Open Label Extension Study to Investigate the Safety of Cannabidiol (GWP42003-P; CBD) in Children and Adults With Inadequately Controlled Dravet or Lennox-Gastaut Syndromes.
Brief Title: An Open Label Extension Study of Cannabidiol (GWP42003-P) in Children and Adults With Dravet or Lennox-Gastaut Syndromes
Acronym: GWPCARE5
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GW Research Ltd (Industry)
Responsible Party: Sponsor
Organization: GWResearch (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GWEP1415; 2014-001834-27 (EudraCT Number)
Record Dates: First submitted 2014-08-21; First posted 2014-08-25 (Estimated); Results first posted 2022-02-03 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Epilepsy; Dravet Syndrome; Lennox-Gastaut Syndrome
Keywords: Cannabidiol; CBD; GWP42003-P; GWPCARE5
MeSH Terms: conditions — Epilepsy; Epilepsies, Myoclonic; Lennox Gastaut Syndrome | interventions — Cannabidiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GWP42003-P (Experimental)
  Interventions: Drug: GWP42003-P

INTERVENTIONS:
Drug: GWP42003-P
  Other Names: Cannabidiol; CBD; Epidiolex/Epidyolex®

SUMMARY:
To investigate the potential antiepileptic effects of cannabidiol (GWP42003-P) in children and adults with Dravet or Lennox-Gastaut syndromes.

DETAILED DESCRIPTION:
This is a multi-center, open-label extension study for participants with Dravet syndrome or Lennox-Gastaut syndrome who have previously participated in double-blind, placebo-controlled clinical studies of GWP42003-P (Core Studies: GWEP1332A [NCT02091206], GWEP1332B [NCT02091375], GWEP1424 [NCT02224703], GWEP1414 [NCT02224560], GWEP1424 [NCT02224703], and GWEP1423 [NCT02224690]). The first participant was enrolled into the open-label extension study after the Data Safety Monitoring Committee reviewed the safety data from Part A of study GWEP1332.

ELIGIBILITY:
Key Inclusion Criteria:

• Participant has completed the treatment phase of their Core Studies: GWEP1332A [NCT02091206], GWEP1332B [NCT02091375], GWEP1424 [NCT02224703], GWEP1414 [NCT02224560], GWEP1424 [NCT02224703], and GWEP1423 [NCT02224690].

Key Exclusion Criteria:

* Participant is currently using or has in the past used recreational or medicinal cannabis, or synthetic cannabinoid-based medications (including Sativex®) within the 3 months prior to study entry other than the investigational medicinal product (IMP) received during the Core Study and are unwilling to abstain for the duration for the study.
* Any history of suicidal behavior or any suicidal ideation of type 4 or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS) at Visit 1.
* Participant has been part of a clinical trial involving an IMP during the inter-study period.
* Female participant is of child bearing potential or male participant's partner is of child bearing potential, unless willing to ensure that they or their partner use highly effective contraception, for example, hormonal contraceptives, intrauterine devices/hormone-releasing systems, bilateral tubal occlusion, vasectomized partner or sexual abstinence, during the study and for 3 months thereafter (however, a male condom should not be used in conjunction with a female condom).
* Participant has significantly impaired hepatic function at the 'End of Treatment' visit of their Core Study or at Visit 1 if re-assessed: i) Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >5 × upper limit of normal (ULN); ii) ALT or AST >3 × ULN and (total bilirubin [TBL] >2 × ULN or international normalized ratio [INR] >1.5); iii) ALT or AST >3 × ULN with the presence of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, and/or eosinophilia (>5%). This criterion must be confirmed prior to entering the study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 681 (Actual)
Dates: Start 2015-06-11 (Actual); Primary Completion 2020-09-24 (Actual); Study Completion 2020-09-24 (Actual)

REFERENCES:
- [Derived] Scheffer IE, Halford JJ, Miller I, Nabbout R, Sanchez-Carpintero R, Shiloh-Malawsky Y, Wong M, Zolnowska M, Checketts D, Dunayevich E, Devinsky O. Add-on cannabidiol in patients with Dravet syndrome: Results of a long-term open-label extension trial. Epilepsia. 2021 Oct;62(10):2505-2517. doi: 10.1111/epi.17036. Epub 2021 Aug 18. PMID 34406656
- [Derived] Patel AD, Mazurkiewicz-Beldzinska M, Chin RF, Gil-Nagel A, Gunning B, Halford JJ, Mitchell W, Scott Perry M, Thiele EA, Weinstock A, Dunayevich E, Checketts D, Devinsky O. Long-term safety and efficacy of add-on cannabidiol in patients with Lennox-Gastaut syndrome: Results of a long-term open-label extension trial. Epilepsia. 2021 Sep;62(9):2228-2239. doi: 10.1111/epi.17000. Epub 2021 Jul 20. PMID 34287833

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who completed the double-blind, placebo-controlled, clinical studies with GWP42003-P (Core Studies: GWEP1332A [NCT02091206], GWEP1332B [NCT02091375], GWEP1424 [NCT02224703], GWEP1414 [NCT02224560], and GWEP1423 [NCT02224690]) were eligible for enrollment.
Groups:
- Dravet Syndrome: Participants with Dravet Syndrome who completed double-blind, placebo-controlled, clinical studies of GWP42003-P (Core Studies: GWEP1332A [NCT02091206], GWEP1332B [NCT02091375], and GWEP1424 [NCT02224703]) were titrated up to 10 to 20 milligrams per kilogram per day (mg/kg/day) GWP42003-P using a recommended titration schedule during the Titration Period. Participants continued at this dose during the Maintenance Period. The maximum dose participants could receive was 30 mg/kg/day.
- Lennox-Gastaut Syndrome: Participants with Lennox-Gastaut Syndrome who completed double-blind, placebo-controlled, clinical studies of GWP42003-P (Core Studies: GWEP1414 [NCT02224560] and GWEP1423 [NCT02224690]) were titrated up to 10 to 20 milligrams per kilogram per day (mg/kg/day) GWP42003-P using a recommended titration schedule during the Titration Period. Participants continued at this dose during the Maintenance Period. The maximum dose participants could receive was 30 mg/kg/day.
Period: Treatment Phase
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Started | 315 | 366
Completed | 170 | 243
Not Completed | 145 | 123
Not completed — Caregiver Asked to Stop Investigational Medicinal Product (IMP) | 0 | 1
Not completed — Started on Other IMP | 1 | 0
Not completed — Participant Discontinued IMP | 0 | 1
Not completed — Lack of Efficacy | 15 | 8
Not completed — Began Commercial Product | 1 | 0
Not completed — Lack of Efficacy per Participant/Caregiver | 3 | 3
Not completed — Met Withdrawal Criteria | 5 | 7
Not completed — Participant Did Not Return for Visits | 0 | 1
Not completed — Continued Compassionate Use | 1 | 0
Not completed — Lack of Efficiency | 2 | 1
Not completed — Participant with Protocol-Excluded Treatment | 0 | 1
Not completed — Participant Moved | 2 | 0
Not completed — Withdrawal by Participant or Parent/Guardian | 62 | 48
Not completed — Refused Medication | 1 | 1
Not completed — Adverse Event | 26 | 38
Not completed — Placed in Group Home | 0 | 1
Not completed — Pursued Other Trials | 1 | 0
Not completed — Withdrawn by the Investigator | 23 | 11
Not completed — Lost to Follow-up | 2 | 1
Period: Taper Phase
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Started | 79 (The number of participants to start the Taper Phase is not equal to the number who completed the Treatment Phase because not all participants tapered IMP.) | 71 (The number of participants to start the Taper Phase is not equal to the number who completed the Treatment Phase because not all participants tapered IMP.)
Completed | 76 | 67
Not Completed | 3 | 4
Not completed — Completed Incorrect Number of Taper Days | 1 | 0
Not completed — Hospitalization/Dose Reduction | 1 | 0
Not completed — Withdrawn by participants or parent/guardian | 0 | 3
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome | Total
Number analyzed (Participants) | 315 | 366 | 681
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.737 (4.4434) | 15.906 (9.5392) | 13.053 (8.2120)
Age, Customized [Count of Participants; unit: Participants]
  Children (2-11 years) | 216 | 157 | 373
  Adolescents (12-17 years) | 90 | 89 | 179
  Adults (18-64 years) | 9 | 120 | 129
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 159 | 168 | 327
  Male | 156 | 198 | 354
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 6 | 10 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 15 | 25
  White | 269 | 325 | 594
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 29 | 16 | 45
Race [Count of Participants; unit: Participants]
  White/Caucasian | 269 | 325 | 594
  Black/African American | 10 | 15 | 25
  American Indian/Alaska Native | 1 | 0 | 1
  Asian | 6 | 10 | 16
  Not Applicable (As per country-specific data protection law. | 15 | 1 | 16
  Caucasian/Asian | 1 | 1 | 2
  Hispanic/Caucasian | 1 | 2 | 3
  White and Black Caribbean | 1 | 0 | 1
  Biracial | 2 | 1 | 3
  Caucasian and African American | 3 | 1 | 4
  Mulatto | 1 | 0 | 1
  North African | 1 | 0 | 1
  South American | 1 | 0 | 1
  Latino | 1 | 5 | 6
  Eurasian | 1 | 0 | 1
  Anglo-Indian | 1 | 0 | 1
  Indian | 0 | 2 | 2
  Unknown | 0 | 2 | 2
  Arab | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE) Occurring in ≥5% of Participants in Any Treatment Group
Description: TEAEs, defined as AEs that started, or worsened in severity or seriousness, following the first dose of investigational medicinal product in this study, are reported. Any AEs that continued from the Core Study (GWEP1332A [NCT02091206], GWEP1332B [NCT02091375], GWEP1424 [NCT02224703], GWEP1414 [NCT02224560], and GWEP1423 [NCT02224690]) were only classified as treatment emergent if they worsened in this study.
Time Frame: up to Week 260
Population: Safety Analysis Set: all participants who received at least 1 dose of investigational medicinal product (IMP).
Measure: Number; unit: participants
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 315 | 366
participants
  Total participants affected by any TEAE | 306 | 353
  Diarrhoea | 135 | 140
  Vomiting | 63 | 107
  Constipation | 20 | 43
  Nausea | 16 | 32
  Pyrexia | 124 | 126
  Fatigue | 39 | 38
  Upper respiratory tract infection | 78 | 104
  Nasopharyngitis | 78 | 58
  Sinusitis | 38 | 49
  Pneumonia | 35 | 51
  Ear infection | 35 | 50
  Influenza | 37 | 45
  Urinary tract infection | 19 | 51
  Pharyngitis streptococcal | 26 | 27
  Gastroenteritis viral | 15 | 30
  Otitis media | 21 | 22
  Bronchitis | 15 | 23
  Viral upper respiratory tract infection | 11 | 20
  Gastroenteritis | 16 | 7
  Fall | 22 | 23
  Laceration | 8 | 35
  Contusion | 15 | 25
  Weight decreased | 21 | 61
  Alanine aminotransferase increased | 37 | 30
  Aspartate aminotransferase increased | 38 | 19
  Gamma-glutamyltransferase increased | 32 | 20
  Decreased appetite | 99 | 93
  Convulsion | 79 | 141
  Somnolence | 87 | 107
  Status epilepticus | 47 | 42
  Lethargy | 21 | 34
  Headache | 18 | 26
  Sedation | 16 | 27
  Drooling | 11 | 21
  Abnormal behaviour | 34 | 23
  Insomnia | 16 | 40
  Irritability | 26 | 29
  Aggression | 20 | 30
  Agitation | 9 | 19
  Cough | 42 | 63
  Nasal congestion | 13 | 46
  Rhinorrhoea | 20 | 19
  Pneumonia aspiration | 4 | 22
  Hypoxia | 2 | 21

2. Primary Outcome: Number of Participants With Clinically Significant Changes in the Indicated Vital Sign Values From the Pre-randomization Baseline of the Core Study at Any Time Post-dose
Description: Clinical significance was determined by the investigator. Pre-randomization Baseline of the Core Study (GWEP1332A [NCT02091206], GWEP1332B [NCT02091375], GWEP1424 [NCT02224703], GWEP1414 [NCT02224560], and GWEP1423 [NCT02224690]) is defined as Baseline of the double-blind, placebo-controlled, clinical studies with GWP42003-P. bpm = beats per minute; DBP = Diastolic Blood Pressure; mmHg = millimeters of mercury; SBP = Systolic Blood Pressure. Data for change from Baseline at pre-randomization of the Core Study are presented; however, the time frame represents the duration for which participants were enrolled in GWEP1415. The only data presented from the Core Studies in this report are the comparison of the Extension Study data with the Baseline data at pre-randomization of the Core Study.
Time Frame: up to Week 260
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 315 | 366
participants
  Sitting SBP < -20 mmHg | 59 | 88
  Sitting SBP > 20 mmHg | 96 | 120
  Sitting DBP < -10 mmHg | 139 | 176
  Sitting DBP > 10 mmHg | 166 | 191
  Pulse Rate < -15 bpm | 176 | 192
  Pulse Rate > 15 bpm | 150 | 179
  Weight ≤ -7 % | 47 | 106
  Weight ≥ 7% | 213 | 223

3. Primary Outcome: Mean Change From the Pre-randomization Baseline of the Core Study to the End of Treatment in Body Mass Index (BMI)
Description: BMI is an estimate of body fat based on body weight divided by height squared. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Pre-randomization Baseline of the Core Study (GWEP1332A [NCT02091206], GWEP1332B [NCT02091375], GWEP1424 [NCT02224703], GWEP1414 [NCT02224560], and GWEP1423 [NCT02224690]) is defined as Baseline of the double-blind, placebo-controlled, clinical studies with GWP42003-P. Data for change from Baseline at pre-randomization of the Core Study are presented; however, the time frame represents the duration for which participants were enrolled in GWEP1415. The only data presented from the Core Studies in this report are the comparison of the Extension Study data with the Baseline data at pre-randomization of the Core Study.
Time Frame: up to Week 260
Population: Safety Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: kilograms per meters squared (kg/m^2)
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 243 | 294
kilograms per meters squared (kg/m^2) | 0.42 (2.701) | 0.05 (5.863)

4. Primary Outcome: Number of Participants With Clinically Significant Electrocardiogram (ECG) Values at the Pre-randomization Baseline of the Core Study and at Any Time Post-dose
Description: Clinical significance was determined by the investigator. Pre-randomization Baseline of the Core Study (GWEP1332A [NCT02091206], GWEP1332B [NCT02091375], GWEP1424 [NCT02224703], GWEP1414 [NCT02224560], and GWEP1423 [NCT02224690]) is defined as Baseline of the double-blind, placebo-controlled, clinical studies with GWP42003-P. msec = milliseconds; QTcB = corrected QT interval with Bazett's correction. The time frame represents the duration for which participants were enrolled in GWEP1415. The only data presented from the Core Studies in this report are the comparison of the Extension Study data with the Baseline data at pre-randomization of the Core Study.
Time Frame: up to Week 260
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 315 | 366
participants
  QTcB > 450 msec, Baseline | 13 | 21
  QTcB > 450 msec, any time post-dose | 62 | 120
  QTcB > 480 msec, Baseline | 2 | 4
  QTcB > 480 msec, any time post-dose | 10 | 40
  QTcB > 500 msec, Baseline | 2 | 2
  QTcB > 500 msec, any time post-dose | 7 | 20

5. Primary Outcome: Number of Participants With the Indicated Responses to Questions Regarding Suicidal Ideation and Behavior Using the Children's Columbia-Suicide Severity Rating Scale (C-SSRS) at Day 1 and at Any Time Post-dose
Description: The C-SSRS questionnaire is a brief, standardized measure that uniquely assesses the essential information (behavior, ideation, lethality, and severity) and distinguishes between suicidal occurrences and non-suicidal self-injury.
Time Frame: up to Week 260
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 315 | 366
participants
  Any suicidality, Day 1 | 1 | 1
  Any suicidality, any time post-dose | 1 | 2
  Suicidal ideation, Day 1 | 0 | 1
  Suicidal ideation, any time post-dose | 1 | 2
  Suicidal behavior, Day 1 | 1 | 0
  Suicidal behavior, any time post-dose | 1 | 0
  Complete suicidality, any time post-dose | 0 | 0

6. Primary Outcome: Mean Cannabis Withdrawal Scale Score at End of Taper (EOT), the Post-Taper Safety Call, and at Safety Follow-up
Description: The Cannabis Withdrawal Scale is a 19-item scale administered to participants (18 years and above), with each item (withdrawal symptom) measured on a 0 to 10 numerical rating scale (0 = Not at all; 5 = Moderately; 10 = Extremely). Total score, calculated as the sum of the 19 item sub-scores ranging from 0-190 are reported. Higher scores indicate more withdrawal symptoms and an increased negative impact to quality of life. The participant or participant's caregiver was asked to record the extent to which each withdrawal symptom was experienced in the last 24 hours and also to rate the negative impact on normal daily activities. L24S = Last 24 Hours Score; NIS = Negative Impact on Normal Daily Activity Score. The End of Treatment visit occurred after a maximum of 260 weeks of treatment. The End of Taper occurred up to 10 days after the End of Treatment visit. The Safety Call and Safety Follow-up occurred 2 and 4 weeks, respectively, after the End of Taper.
Time Frame: up to Week 260
Population: Safety Analysis Set. Only participants (18 years and above) with available Cannabis Withdrawal Scale score were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 315 | 366
scores on a scale
  L24S, End of Taper: number analyzed (Participants) | 5 | 11
  L24S, End of Taper | 9.8 (10.64) | 4.9 (14.00)
  L24S, Post-Taper Safety Call: number analyzed (Participants) | 5 | 8
  L24S, Post-Taper Safety Call | 3.4 (4.72) | 0.0 (0.00)
  L24S, Safety Follow-Up: number analyzed (Participants) | 5 | 11
  L24S, Safety Follow-Up | 2.4 (3.36) | 4.9 (12.27)
  NIS, End of Taper: number analyzed (Participants) | 6 | 18
  NIS, End of Taper | 9.5 (12.03) | 5.1 (10.96)
  NIS, Post-Taper Safety Call: number analyzed (Participants) | 3 | 13
  NIS, Post-Taper Safety Call | 16.3 (3.79) | 1.2 (3.00)
  NIS, Safety Follow-Up: number analyzed (Participants) | 3 | 10
  NIS, Safety Follow-Up | 5.3 (9.24) | 1.8 (3.82)

7. Primary Outcome: Mean Pediatric Cannabinoid Withdrawal Scale (PCWS) Score at the End of Treatment, the End of Taper, the Post-Taper Safety Call, and at Safety Follow-up
Description: The PCWS was administered to participants aged 4 to 17 (inclusive) that was developed from the 19-item validated CWS (adults) to assess mood, behavioral, and physical symptoms associated with cannabis. The total score, calculated as the sum of 10 items (rated on a 4-point scale: 0 = none; 1 = a little bit; 2 = quite a bit; 3 = a lot) ranging from 0-30 are reported. Higher scores indicate more withdrawal symptoms and an increased negative impact to quality of life. The End of Treatment visit occurred after a maximum of 260 weeks of treatment. The participant or participant's caregiver was asked to record the extent to which each withdrawal symptom was experienced in the last 24 hours and also to rate the negative impact on normal daily activities. The End of Taper occurred up to 10 days after the End of Treatment visit. The Safety Call and Safety Follow-up occurred 2 and 4 weeks, respectively, after the End of Taper.
Time Frame: up to Week 260
Population: Safety Analysis Set. Only participants (4 to 17 years) with available Pediatric Cannabis Withdrawal Scale score were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 74 | 46
scores on a scale
  End of Treatment: number analyzed (Participants) | 1 | 1
  End of Treatment | 4.0 (NA) — Only 1 participant was analyzed so SD could not be evaluated. | 6.0 (NA) — Only 1 participant was analyzed so SD could not be evaluated.
  End of Taper | 2.9 (3.77) | 2.1 (2.78)
  Post-Taper Safety Call: number analyzed (Participants) | 55 | 25
  Post-Taper Safety Call | 2.4 (3.50) | 2.0 (2.72)
  Safety Follow-Up: number analyzed (Participants) | 68 | 34
  Safety Follow-Up | 1.9 (2.72) | 1.8 (2.28)

8. Primary Outcome: Mean Change From the Pre-randomization Baseline of the Core Study to the End of Treatment in Red Blood Cells (RBCs) Values
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Pre-randomization Baseline of the Core Study (GWEP1332A [NCT02091206], GWEP1332B [NCT02091375], GWEP1424 [NCT02224703], GWEP1414 [NCT02224560], and GWEP1423 [NCT02224690]) is defined as Baseline of the double-blind, placebo-controlled, clinical studies with GWP42003-P. Data for change from Baseline at pre-randomization of the Core Study are presented; however, the time frame represents the duration for which participants were enrolled in GWEP1415. The only data presented from the Core Studies in this report are the comparison of the Extension Study data with the Baseline data at pre-randomization of the Core Study.
Time Frame: up to Week 260
Population: Safety Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: 10^12 cells per Liter (L)
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 268 | 307
10^12 cells per Liter (L) | -0.068 (0.3297) | -0.059 (0.3424)

9. Primary Outcome: Mean Change From the Pre-randomization Baseline of the Core Study to the End of Treatment in Hemoglobin Levels
Description: as for outcome 8
Time Frame: up to Week 260
Population: Safety Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: grams per Liter (g/L)
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 268 | 307
grams per Liter (g/L) | -1.6 (9.08) | -2.4 (11.14)

10. Primary Outcome: Mean Change From the Pre-randomization Baseline of the Core Study to the End of Treatment in Hematocrit Values
Description: as for outcome 8
Time Frame: up to Week 260
Population: Safety Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of RBCs in whole blood (L/L)
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 268 | 307
percentage of RBCs in whole blood (L/L) | -0.0105 (0.02938) | -0.0110 (0.02983)

11. Primary Outcome: Mean Change From the Pre-randomization Baseline of the Core Study to the End of Treatment in Erythrocyte Mean Corpuscular Volume
Description: as for outcome 8
Time Frame: up to Week 260
Population: Safety Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: femtoliters (fL)
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 268 | 307
femtoliters (fL) | -1.0 (5.10) | -1.3 (5.01)

12. Primary Outcome: Mean Change From the Pre-randomization Baseline of the Core Study to the End of Treatment in Erythrocyte Mean Corpuscular Hemoglobin
Description: as for outcome 8
Time Frame: up to Week 260
Population: Safety Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: picograms (pg)
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 268 | 307
picograms (pg) | 0.10 (1.482) | -0.15 (1.926)

13. Primary Outcome: Mean Change From the Pre-randomization Baseline of the Core Study to the End of Treatment in Platelets, White Blood Cells, Basophils, Eosinophils, Lymphocytes, Monocytes, and Neutrophils
Description: as for outcome 8
Time Frame: up to Week 260
Population: Safety Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 315 | 366
10^9 cells/L
  Platelets: number analyzed (Participants) | 266 | 304
  Platelets | 5.4 (64.84) | 5.0 (70.47)
  White blood cells: number analyzed (Participants) | 268 | 307
  White blood cells | -0.52 (2.531) | -0.09 (2.052)
  Basophils: number analyzed (Participants) | 268 | 305
  Basophils | 0.00 (0.041) | 0.01 (0.040)
  Eosinophils: number analyzed (Participants) | 268 | 305
  Eosinophils | -0.02 (0.159) | -0.02 (0.165)
  Lymphocytes: number analyzed (Participants) | 268 | 305
  Lymphocytes | -0.31 (0.988) | -0.14 (0.778)
  Monocytes: number analyzed (Participants) | 268 | 305
  Monocytes | -0.05 (0.276) | 0.01 (0.245)
  Neutrophils: number analyzed (Participants) | 268 | 305
  Neutrophils | -0.16 (2.041) | 0.05 (1.878)

14. Primary Outcome: Mean Change From the Pre-randomization Baseline of the Core Study to the End of Treatment in the Percentage of Basophils, Eosinophils, Lymphocytes, Monocytes, and Neutrophils in White Blood Cells (WBCs)
Description: as for outcome 8
Time Frame: up to Week 260
Population: Safety Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage in WBCs
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 268 | 305
percentage in WBCs
  Basophils/WBCs | 0.08 (0.284) | 0.12 (0.287)
  Eosinophils/WBCs | -0.10 (2.064) | -0.24 (2.104)
  Lymphocytes/WBCs | -1.32 (12.396) | -1.32 (11.193)
  Monocytes/WBCs | -0.05 (3.125) | 0.18 (2.600)
  Neutrophils/WBCs | 1.47 (12.982) | 1.27 (12.245)

15. Primary Outcome: Mean Change From the Pre-randomization Baseline of the Core Study to the End of Treatment in Sodium, Potassium, Blood Urea Nitrogen, Glucose, Calcium, and High-Density Lipoprotein (HDL) Cholesterol
Description: as for outcome 8
Time Frame: up to week 260
Population: Safety Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: millimoles per Liter (mmol/L)
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 315 | 366
millimoles per Liter (mmol/L)
  Sodium: number analyzed (Participants) | 277 | 311
  Sodium | -0.4 (3.25) | -0.8 (2.70)
  Potassium: number analyzed (Participants) | 274 | 307
  Potassium | -0.06 (0.372) | -0.08 (0.407)
  Blood urea nitrogen: number analyzed (Participants) | 276 | 309
  Blood urea nitrogen | -0.08 (1.571) | 0.00 (1.555)
  Glucose: number analyzed (Participants) | 275 | 307
  Glucose | -0.06 (1.026) | 0.06 (1.288)
  Calcium: number analyzed (Participants) | 277 | 311
  Calcium | -0.050 (0.1148) | -0.054 (0.1218)
  HDL cholesterol: number analyzed (Participants) | 277 | 311
  HDL cholesterol | 0.06 (0.372) | 0.12 (0.320)

16. Primary Outcome: Mean Change From the Pre-randomization Baseline of the Core Study to the End of Treatment in Creatinine (Jaffe), Creatinine (Enzymatic), and Bilirubin
Description: as for outcome 8
Time Frame: up to Week 260
Population: Safety Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: micromoles per Liter (µmol/L)
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 315 | 366
micromoles per Liter (µmol/L)
  Creatinine, Jaffe: number analyzed (Participants) | 268 | 311
  Creatinine, Jaffe | 7.0 (9.32) | 7.1 (10.86)
  Creatinine, enzymatic: number analyzed (Participants) | 148 | 140
  Creatinine, enzymatic | 3.8 (8.83) | 4.0 (9.44)
  Bilirubin: number analyzed (Participants) | 276 | 309
  Bilirubin | 0.48 (2.339) | 0.45 (2.626)

17. Primary Outcome: Mean Change From the Pre-randomization Baseline of the Core Study to the End of Treatment in Creatinine Clearance (Schwartz) and Creatinine Clearance (Cockcroft-Gault)
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Pre-randomization Baseline of the Core Study (GWEP1332A [NCT02091206], GWEP1332B [NCT02091375], GWEP1424 [NCT02224703], GWEP1414 [NCT02224560], and GWEP1423 [NCT02224690]) is defined as Baseline of the double-blind, placebo-controlled, clinical studies with GWP42003-P. mL/min/1.73 m^2 = millilitres per minute per 1.73 meters squared. Data for change from Baseline at pre-randomization of the Core Study are presented; however, the time frame represents the duration for which participants were enrolled in GWEP1415. The only data presented from the Core Studies in this report are the comparison of the Extension Study data with the Baseline data at pre-randomization of the Core Study.
Time Frame: up to Week 260
Population: Safety Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 315 | 366
mL/min/1.73 m^2
  Creatinine Clearance, Schwartz,: number analyzed (Participants) | 247 | 185
  Creatinine Clearance, Schwartz, | 0.3 (4.41) | 0.0 (0.00)
  Creatinine Clearance, Cockcroft-Gault: number analyzed (Participants) | 7 | 103
  Creatinine Clearance, Cockcroft-Gault | 0.0 (0.00) | -0.6 (5.94)

18. Primary Outcome: Mean Change From the Pre-randomization Baseline of the Core Study to the End of Treatment in Alkaline Phosphatase, Aspartate Aminotransferase, Alanine Aminotransferase, and Gamma Glutamyl Transferase
Description: as for outcome 8
Time Frame: up to Week 260
Population: Safety Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Units/L
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 315 | 366
Units/L
  Alkaline phosphatase: number analyzed (Participants) | 277 | 311
  Alkaline phosphatase | -40.9 (88.18) | -40.1 (73.62)
  Aspartate aminotransferase: number analyzed (Participants) | 274 | 308
  Aspartate aminotransferase | 4.0 (26.14) | 2.8 (26.62)
  Alanine aminotransferase: number analyzed (Participants) | 275 | 308
  Alanine aminotransferase | 7.0 (39.24) | 9.5 (43.96)
  Gamma glutamyl transferase: number analyzed (Participants) | 276 | 309
  Gamma glutamyl transferase | 8.7 (42.35) | 4.9 (45.65)

19. Primary Outcome: Mean Change From the Pre-randomization Baseline of the Core Study to the End of Treatment in Albumin and Protein
Description: as for outcome 8
Time Frame: up to Week 260
Population: Safety Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: grams (g)/L
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 315 | 366
grams (g)/L
  Albumin: number analyzed (Participants) | 277 | 311
  Albumin | -0.2 (3.43) | -0.9 (3.31)
  Protein: number analyzed (Participants) | 277 | 311
  Protein | -1.2 (5.83) | -2.0 (5.75)

20. Primary Outcome: Mean Change From the Pre-randomization Baseline of the Core Study to the End of Treatment in Prolactin
Description: as for outcome 8
Time Frame: up to Week 260
Population: Safety Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: µInternational Units/millilitre (µIU/mL)
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 276 | 309
µInternational Units/millilitre (µIU/mL) | 0.43 (132.613) | 10.43 (230.439)

21. Primary Outcome: Mean Change From the Pre-randomization Baseline of the Core Study to the End of Treatment in Prothrombin Time
Description: as for outcome 8
Time Frame: up to Week 260
Population: Safety Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 256 | 282
seconds | -0.08 (0.740) | -0.09 (0.706)

22. Primary Outcome: Mean Change From the Pre-randomization Baseline of the Core Study to the End of Treatment in Prothrombin International Normalized Ratio
Description: as for outcome 8
Time Frame: up to Week 260
Population: Safety Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 256 | 282
ratio | -0.012 (0.0784) | -0.010 (0.0736)

23. Primary Outcome: Mean Change From the Pre-randomization Baseline of the Core Study to the End of Treatment in Insulin-like Growth Factor-1 (IGF-1) Levels
Description: IGF-1 levels in serum were analyzed as part of the clinical laboratory testing in participants. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Pre-randomization Baseline of the Core Study (GWEP1332A [NCT02091206], GWEP1332B [NCT02091375], GWEP1424 [NCT02224703], GWEP1414 [NCT02224560], and GWEP1423 [NCT02224690]) is defined as Baseline of the double-blind, placebo-controlled, clinical studies with GWP42003-P. Data for change from Baseline at pre-randomization of the Core Study are presented; however, the time frame represents the duration for which participants were enrolled in GWEP1415. The only data presented from the Core Studies in this report are the comparison of the Extension Study data with the Baseline data at pre-randomization of the Core Study.
Time Frame: up to Week 260
Population: Safety Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: nanomoles (nmol)/L
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 69 | 142
nanomoles (nmol)/L | -0.28 (12.701) | 1.10 (15.970)

24. Primary Outcome: Mean Subject/Caregiver Global Impression of Change (S/CGIC) Score
Description: The S/CGIC allows participants and caregivers to rate the participant's overall condition on a scale of 1 to 7 (1 = Very Much Improved, and 7 = Very Much Worse). The combined caregiver and participant summary used either the caregiver or participant version if only one version was completed, or the caregiver version when both the caregiver and participant versions were completed. The only data presented from the Core Studies in this report are the comparison of the Extension Study data with the Baseline data at pre-randomization of the Core Study.
Time Frame: Baseline; up to Week 260
Population: Safety Analysis Set. Only those participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 315 | 366
Scores on a scale | 3.0 (1.47) | 2.8 (1.38)

25. Primary Outcome: Percent Change From the Pre-randomization Baseline of the Core Study to the End of Treatment in Total Seizure Frequency
Description: Total seizures included the sum of all seizures (tonic-clonic, tonic, atonic, clonic, myoclonic, countable partial, other partial, and absence seizures) recorded by the participant or caregiver. Change from Baseline was calculated as the percentage change from Baseline for each 12-week period. Pre-randomization Baseline of the Core Study (GWEP1332A [NCT02091206], GWEP1332B [NCT02091375], GWEP1424 [NCT02224703], GWEP1414 [NCT02224560], and GWEP1423 [NCT02224690]) is defined as Baseline of the double-blind, placebo-controlled, clinical studies with GWP42003-P. The only data presented from the Core Studies in this report are the comparison of the Extension Study data with the Baseline data at pre-randomization of the Core Study. "Last 12 weeks" is equal to the last 12 weeks' data for each participant irrespective of time in study.
Time Frame: Baseline; Week 49 to 60, Week 97 to 108, Week 145 to 156, Week 205 to 216, Week 253 to 264, and Last 12 Weeks
Population: Safety Analysis Set. Only participants with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: percentage change
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 315 | 366
percentage change
  Week 49 to 60: number analyzed (Participants) | 174 | 283
  Week 49 to 60 | -65.8 [-86.9 to -19.8] | -58.9 [-84.6 to -26.9]
  Week 97 to 108: number analyzed (Participants) | 111 | 228
  Week 97 to 108 | -71.3 [-93.8 to -14.3] | -66.4 [-86.2 to -34.2]
  Week 145 to 156: number analyzed (Participants) | 67 | 202
  Week 145 to 156 | -79.8 [-97.6 to -5.3] | -65.3 [-88.2 to -32.0]
  Week 205 to 216: number analyzed (Participants) | 9 | 15
  Week 205 to 216 | -81.5 [-93.0 to -73.3] | -78.4 [-94.3 to -52.4]
  Week 253 to 264: number analyzed (Participants) | 3 | 0
  Week 253 to 264 | -70.0 [-83.1 to 178.6] |
  Last 12 weeks: number analyzed (Participants) | 290 | 363
  Last 12 weeks | -55.2 [-84.0 to 2.9] | -51.9 [-84.7 to -13.3]

26. Primary Outcome: Percent Change From the Pre-randomization Baseline of the Core Study to the End of Treatment in Drop Seizure Frequency in Participants With Lennox-Gastaut Syndrome
Description: Drop seizures are defined as the subset of tonic-clonic, tonic, or atonic seizures. Change from Baseline was calculated as the percentage change from Baseline for each 12-week period. Pre-randomization Baseline of the Core Study (GWEP1332A [NCT02091206], GWEP1332B [NCT02091375], GWEP1424 [NCT02224703], GWEP1414 [NCT02224560], and GWEP1423 [NCT02224690]) is defined as Baseline of the double-blind, placebo-controlled, clinical studies with GWP42003-P. Data for change from Baseline at pre-randomization of the Core Study are presented; however, the time frame represents the duration for which participants were enrolled in GWEP1415. The only data presented from the Core Studies in this report are the comparison of the Extension Study data with the Baseline data at pre-randomization of the Core Study. The outcome was reported for Lennox-Gastaut Syndrome participants only. "Last 12 weeks" is equal to the last 12 weeks' data for each participant irrespective of time in study.
Time Frame: Baseline; Week 49 to 60, Week 97 to 108, Week 145 to 156, Week 205 to 216, and Last 12 Weeks
Population: Safety Analysis Set. Only participants with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: percentage change
Arm/Group | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 366
percentage change
  Week 49 to 60: number analyzed (Participants) | 283
  Week 49 to 60 | -59.4 [-85.9 to -22.5]
  Week 97 to 108: number analyzed (Participants) | 228
  Week 97 to 108 | -69.4 [-91.3 to -27.9]
  Week 145 to 156: number analyzed (Participants) | 202
  Week 145 to 156 | -70.8 [-90.8 to -37.5]
  Week 205 to 216: number analyzed (Participants) | 15
  Week 205 to 216 | -68.7 [-98.8 to -33.3]
  Last 12 weeks: number analyzed (Participants) | 363
  Last 12 weeks | -59.4 [-87.1 to -15.4]

27. Primary Outcome: Percent Change From the Pre-randomization Baseline of the Core Study to the End of Treatment in Convulsive Seizure Frequency in Participants With Dravet Syndrome
Description: Convulsive seizures are defined as tonic-clonic, tonic, clonic, or atonic seizures. Change from Baseline was calculated as the percentage change from Baseline for each 12-week period. Pre-randomization Baseline of the Core Study (GWEP1332A [NCT02091206], GWEP1332B [NCT02091375], GWEP1424 [NCT02224703], GWEP1414 [NCT02224560], and GWEP1423 [NCT02224690]) is defined as Baseline of the double-blind, placebo-controlled, clinical studies with GWP42003-P. Data for change from Baseline at pre-randomization of the Core Study are presented; however, the time frame represents the duration for which participants were enrolled in GWEP1415. The only data presented from the Core Studies in this report are the comparison of the Extension Study data with the Baseline data at pre-randomization of the Core Study. The outcome was reported for Dravet Syndrome participants only. "Last 12 weeks" is equal to the last 12 weeks' data for each participant irrespective of time in study.
Time Frame: Baseline; Week 49 to 60, Week 97 to 108, Week 145 to 156, Week 205 to 216, Week 253 to 264, and Last 12 Weeks
Population: Safety Analysis Set. Only participants with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: percentage change
Arm/Group | Dravet Syndrome
Number analyzed (Participants) | 315
percentage change
  Week 49 to 60: number analyzed (Participants) | 174
  Week 49 to 60 | -52.9 [-81.8 to -6.5]
  Week 97 to 108: number analyzed (Participants) | 111
  Week 97 to 108 | -64.3 [-91.7 to -22.2]
  Week 145 to 156: number analyzed (Participants) | 67
  Week 145 to 156 | -69.4 [-96.1 to -24.1]
  Week 205 to 216: number analyzed (Participants) | 9
  Week 205 to 216 | -72.3 [-77.4 to -55.6]
  Week 253 to 264: number analyzed (Participants) | 3
  Week 253 to 264 | -55.6 [-70.0 to 91.7]
  Last 12 weeks: number analyzed (Participants) | 289
  Last 12 weeks | -40.0 [-77.8 to 6.7]

28. Primary Outcome: Number of Participants With Convulsive and Non-convulsive Seizures Greater Than 30 Minutes in Duration (Status Epilepticus)
Description: Status epilepticus is defined as any seizure lasting for 30 minutes or longer. The number of convulsive seizures greater than 30 minutes in duration and the number of non-convulsive seizures greater than 30 minutes in duration were collected weekly. The only data presented from the Core Studies in this report are the comparison of the Extension Study data with the Baseline data at pre-randomization of the Core Study. mins = minutes. "Last 12 weeks" is equal to the last 12 weeks' data for each participant irrespective of time in study.
Time Frame: Baseline; At last 12 weeks
Population: Safety Analysis Set. Only participants with available data are analyzed.
Measure: Number; unit: participants
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 315 | 366
participants
  Convulsive SE: Over the 4-week Baseline; Yes | 14 | 14
  Convulsive SE: Last 12 Weeks; Yes | 13 | 7
  Convulsive SE: Over the 4-week Baseline; No | 277 | 352
  Convulsive SE: Last 12 Weeks; No | 277 | 356
  Non-Convulsive SE: Over the 4-week Baseline; Yes | 21 | 17
  Non-Convulsive SE: Last 12 Weeks; Yes | 14 | 11
  Non-Convulsive SE: Over the 4-week Baseline; No | 270 | 349
  Non-Convulsive SE: Last 12 Weeks; No | 276 | 352

29. Secondary Outcome: Mean Change From the Pre-randomization Baseline of the Core Study to the End of Treatment in Quality of Life in Childhood Epilepsy (QOLCE) Scores
Description: The QOLCE is a parent-reported questionnaire that evaluates health-related QOL in children aged 2-18 years old. It contains 76 items with 16 subscales covering 7 domains (physical activities, social activities, cognition, emotional well-being, behavior, general health, and general QOL). All items in the questionnaire are rated on a 5-point or 6-point categorical scale. Based on the responses to the items in each domain, scores for 16 subscales are derived. Score range from 0 to 100. Higher score indicate highest level of functioning. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Pre-randomization Baseline of the Core Study is defined as the Baseline of the double-blind, placebo-controlled, clinical studies with GWP42003-P. The only data presented from the Core Studies in this report are the comparison of the Extension Study data with the Baseline data at pre-randomization of the Core Study.
Time Frame: Baseline; up to Week 260
Population: Safety Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 169 | 118
Scores on a scale | 3.7 (14.61) | 6.0 (13.87)

30. Secondary Outcome: Mean Change From the Pre-randomization Baseline of the Core Study to the End of Treatment QOL in Epilepsy Scores (QOLIE-31-P) in Participants With Lennox-Gastaut Syndrome
Description: The QOLIE-31-P is a survey of health-related QOL for adults with epilepsy. It is comprised of 38 questions about health daily activities and evaluates how much distress the participant feels about problems and worries related to epilepsy. The questionnaire consists of 7 subscales (energy, mood, daily activities, cognition, medication effects, seizure worry, and overall QOL). Scores range from 0 to 100. Higher scores indicate better QOL. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Pre-randomization Baseline of the Core Study is defined as Baseline of the double-blind, placebo-controlled, clinical studies with GWP42003-P. The only data presented from the Core Studies in this report are the comparison of the Extension Study data with the Baseline data at pre-randomization of the Core Study. The outcome was reported for Lennox-Gastaut Syndrome participants only.
Time Frame: Baseline; up to Week 260
Population: Safety Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 38
Scores on a scale | 1.3 (16.33)

31. Secondary Outcome: Mean Change From the Pre-randomization Baseline of the Core Study to the End of Treatment in Vineland Adaptive Behavior Scale, Second Edition (Vineland-II) Scores
Description: The Vineland-II is an individually administered instrument for assessing adaptive behaviors. It consists of 4 adaptive behavior domains (1 = low; 5 = high) and a maladaptive behavior domain (1 = clinically significant; 3 = average), and an overall Adaptive Behavior Composite Score. Standard scores (population mean = 100, SD = 15, range = 20 to 160) are produced for the domain and composite scores, and scaled scores (called v-scale scores, with a population mean = 15, SD = 3, range = 1 to 24) are produced for the subscale scores. Higher scores indicate better functioning.
  Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Pre-randomization Baseline of the Core Study is defined as Baseline of the double-blind, placebo-controlled, clinical studies with GWP42003-P. The only data presented from the Core Studies in this report are the comparison of the Extension Study data with the Baseline data at pre-randomization of the Core Study.
Time Frame: Baseline; up to Week 260
Population: Safety Analysis Set. Only those participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 315 | 366
Scores on a scale
  Communication: Receptive Subdomain v-Scale Score: number analyzed (Participants) | 93 | 109
  Communication: Receptive Subdomain v-Scale Score | -0.4 (2.12) | -0.5 (2.76)
  Communication: Expressive Subdomain v-Scale Score: number analyzed (Participants) | 96 | 124
  Communication: Expressive Subdomain v-Scale Score | -0.8 (1.65) | -0.3 (2.20)
  Communication: Written Subdomain v-Scale Score: number analyzed (Participants) | 133 | 187
  Communication: Written Subdomain v-Scale Score | -1.1 (1.80) | -0.7 (1.80)
  Communication Domain Standard Score: number analyzed (Participants) | 82 | 105
  Communication Domain Standard Score | -3.2 (8.75) | -1.6 (13.50)
  Daily Living Skills: Personal Subdomain v-Scale Score: number analyzed (Participants) | 113 | 164
  Daily Living Skills: Personal Subdomain v-Scale Score | -1.0 (1.92) | -0.8 (2.05)
  Daily Living Skills: Domestic Subdomain v-Scale Score: number analyzed (Participants) | 114 | 175
  Daily Living Skills: Domestic Subdomain v-Scale Score | -0.8 (2.04) | -1.0 (1.32)
  Daily Living Skills: Community Subdomain v-Scale Score: number analyzed (Participants) | 109 | 165
  Daily Living Skills: Community Subdomain v-Scale Score | -0.9 (2.75) | -0.8 (1.49)
  Daily Living Skills Domain Standard Score: number analyzed (Participants) | 91 | 144
  Daily Living Skills Domain Standard Score | -5.0 (9.68) | -3.9 (8.40)
  Socialization: Interpersonal Relationships Subdomain v-Scale Score: number analyzed (Participants) | 84 | 145
  Socialization: Interpersonal Relationships Subdomain v-Scale Score | -0.7 (1.66) | -0.6 (2.17)
  Socialization: Play and Leisure Time Subdomain v-Scale Score: number analyzed (Participants) | 89 | 142
  Socialization: Play and Leisure Time Subdomain v-Scale Score | -0.9 (2.29) | -0.4 (2.22)
  Socialization: Coping Skills Subdomain v-Scale Score: number analyzed (Participants) | 129 | 187
  Socialization: Coping Skills Subdomain v-Scale Score | -0.7 (2.24) | -0.5 (1.85)
  Socialization Domain Standard Score: number analyzed (Participants) | 76 | 123
  Socialization Domain Standard Score | -3.3 (9.38) | -3.4 (11.29)
  Motor Skills: Gross Subdomain v-Scale Score: number analyzed (Participants) | 105 | 146
  Motor Skills: Gross Subdomain v-Scale Score | -0.2 (1.64) | -0.3 (1.88)
  Motor Skills: Fine Subdomain v-Scale Score: number analyzed (Participants) | 108 | 147
  Motor Skills: Fine Subdomain v-Scale Score | -0.3 (1.99) | -0.4 (2.19)
  Motor Skills Domain Standard Score: number analyzed (Participants) | 94 | 127
  Motor Skills Domain Standard Score | -0.7 (9.62) | -1.9 (10.23)
  Adaptive Behavior Composite Standard Score: number analyzed (Participants) | 66 | 94
  Adaptive Behavior Composite Standard Score | -3.4 (8.09) | -2.5 (10.07)
  Maladaptive Behavior Index: Internalizing Subdomain v-Scale Score: number analyzed (Participants) | 168 | 193
  Maladaptive Behavior Index: Internalizing Subdomain v-Scale Score | -0.1 (2.28) | -0.1 (2.64)
  Maladaptive Behavior Index: Externalizing Subdomain v-Scale Score: number analyzed (Participants) | 158 | 193
  Maladaptive Behavior Index: Externalizing Subdomain v-Scale Score | -0.3 (2.22) | -0.1 (2.12)
  Maladaptive Behavior Index v-Scale Score: number analyzed (Participants) | 132 | 143
  Maladaptive Behavior Index v-Scale Score | -0.3 (1.92) | -0.3 (2.09)

32. Secondary Outcome: Number of Participants With Inpatient Hospitalizations Due to Epilepsy Since the Previous Visit
Description: Inpatient hospitalizations due to epilepsy were recorded by the investigator. The timing of the "End of Treatment" varied per participant based on when the participant discontinued IMP.
Time Frame: Week 48, 104, 156, 208, and End of Treatment (up to Week 260 based on when the participant discontinued treatment)
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 315 | 366
Participants
  Week 48 | 5 | 9
  Week 104 | 4 | 9
  Week 156 | 3 | 0
  Week 208 | 0 | 0
  End of Treatment | 16 | 17

33. Secondary Outcome: Number of Treatment Responders With Greater Than or Equal to 50% Reduction in Total Seizures
Description: Total seizures included the sum of all seizures (tonic-clonic, tonic, atonic, clonic, myoclonic, countable partial, other partial, and absence seizures) recorded by the participant or caregiver.
Time Frame: Baseline; Week 49 to 60, Week 97 to 108, Week 145 to 156, Week 205 to 216, Week 253 to 264, and Last 12 Weeks
Population: Safety Analysis Set. Only participants with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 315 | 366
Participants
  Week 49 to 60: number analyzed (Participants) | 291 | 366
  Week 49 to 60 | 108 | 169
  Week 97 to 108: number analyzed (Participants) | 291 | 366
  Week 97 to 108 | 73 | 148
  Week 145 to 156: number analyzed (Participants) | 291 | 366
  Week 145 to 156 | 48 | 128
  Week 205 to 216: number analyzed (Participants) | 291 | 366
  Week 205 to 216 | 7 | 12
  Week 253 to 264: number analyzed (Participants) | 291 | 0
  Week 253 to 264 | 2 |
  Last 12 Weeks: number analyzed (Participants) | 291 | 366
  Last 12 Weeks | 153 | 188

34. Secondary Outcome: Number of Participants With Changes in the Average Duration of Seizure Subtypes as Assessed by the Participant/Caregiver Global Impression of Change in Seizure Duration (S/CGICSD)
Description: The SGICSD and CGICSD are comprised of the following questions rated on a 3-point scale for each seizure type. The CGICSD score is used to assess the average duration of the participant's seizures (comparing their condition now to their condition before treatment) and the SGICSD score is used to assess the average duration of seizures (comparing condition now to condition before treatment). Scores range from 1 to 3 (1 = Decrease in average duration; 3 = Increase in average duration).
Time Frame: Up to Week 260
Population: Safety Analysis Set. Only participants with available data are analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 291 | 366
Participants
  Tonic-Clonic Seizures; End of Treatment: number analyzed (Participants) | 106 | 125
  Tonic-Clonic Seizures; End of Treatment: Decrease in average duration | 89 | 101
  Tonic-Clonic Seizures; End of Treatment: Increase in average duration | 17 | 24
  Tonic Seizures; End of Treatment: number analyzed (Participants) | 47 | 150
  Tonic Seizures; End of Treatment: Decrease in average duration | 39 | 132
  Tonic Seizures; End of Treatment: Increase in average duration | 8 | 18
  Clonic Seizures; End of Treatment: number analyzed (Participants) | 45 | 41
  Clonic Seizures; End of Treatment: Decrease in average duration | 41 | 38
  Clonic Seizures; End of Treatment: Increase in average duration | 4 | 3
  Atonic Seizures; End of Treatment: number analyzed (Participants) | 32 | 108
  Atonic Seizures; End of Treatment: Decrease in average duration | 26 | 98
  Atonic Seizures; End of Treatment: Increase in average duration | 6 | 10
  Myoclonic Seizures; End of Treatment: number analyzed (Participants) | 62 | 76
  Myoclonic Seizures; End of Treatment: Decrease in average duration | 48 | 72
  Myoclonic Seizures; End of Treatment: Increase in average duration | 14 | 4
  Countable Partial Seizures; End of Treatment: number analyzed (Participants) | 42 | 46
  Countable Partial Seizures; End of Treatment: Decrease in average duration | 34 | 41
  Countable Partial Seizures; End of Treatment: Increase in average duration | 8 | 5
  Other Partial Seizures; End of Treatment: number analyzed (Participants) | 31 | 29
  Other Partial Seizures; End of Treatment: Decrease in average duration | 25 | 29
  Other Partial Seizures; End of Treatment: Increase in average duration | 6 | 0
  Absence Seizures; End of Treatment: number analyzed (Participants) | 51 | 86
  Absence Seizures; End of Treatment: Decrease in average duration | 42 | 83
  Absence Seizures; End of Treatment: Increase in average duration | 9 | 3

35. Secondary Outcome: Mean Change From the Pre-randomization Baseline of the Core Study to the End of Treatment in Delis-Kaplan Executive Function System (D-KEFS) Visual Scanning Completion Time Scaled Score
Description: D-KEFS Visual Scanning Completion Time Scale was used to measure visual attention and processing speed. The cognitive assessment battery items are age-specific, used to measure a variety of functions for both children and adults. The items were administered by an experienced psychometrician to a sub-group of sites that had the expertise to conduct the test. The raw score i.e., total time in seconds for completing the visual scanning trial was measured in the range of 0-150; higher scores indicated worse functioning. The raw score was normed with a referenced score to convert into a scaled score (i.e., score on a scale) ranging from 1-19; higher scores indicated better functioning. Change from the pre-randomization Baseline of the core study to the End of Treatment are reported as score on a scale. Negative values indicate worsening and positive values indicate improvement in cognitive function.
Time Frame: Baseline; up to Week 260
Population: ITT Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 2 | 3
Score on a scale | 0.00 (0.00) | -0.33 (0.577)

36. Secondary Outcome: Mean Change From the Pre-randomization Baseline of the Core Study to the End of Treatment in D-KEFS Number Sequencing Completion Time Scaled Score
Description: D-KEFS Number Sequencing Completion Time Scale was used to measure processing speed. The raw score i.e., total time in seconds for completing the number sequencing trial was measured in the range of 0-150; higher scores indicated worse functioning. The raw score was normed with a referenced score to convert into a scaled score (i.e., score on a scale) ranging from 1-19; higher scores indicated better processing speed. Change from the pre-randomization Baseline of the core study to the End of Treatment are reported as score on a scale. Negative values indicate worsening and positive values indicate improvement in processing speed. The only data presented from the Core Studies in this report are the comparison of the Extension Study data with the Baseline data at pre-randomization of the Core Study.
Time Frame: Baseline; up to Week 260
Population: ITT Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 2 | 2
Score on a scale | 0.00 (0.00) | 0.00 (0.00)

37. Secondary Outcome: Mean Change From the Pre-randomization Baseline of the Core Study to the End of Treatment in D-KEFS Letter Sequencing Completion Time Scaled Score
Description: D-KEFS Letter Sequencing Completion Time Scaled was used to measure processing speed. The raw score i.e., total time in seconds for completing the letter sequencing trial was measured in the range of 0-150; higher scores indicated worse functioning. The raw score was normed with a referenced score to calculate a scaled score (i.e., score on a scale) ranging from 1-19; higher scores indicated better processing speed. Change from the pre-randomization Baseline of the core study to the End of Treatment are reported as score on a scale. Negative values indicate worsening and positive values indicate improvement in processing speed. The only data presented from the Core Studies in this report are the comparison of the Extension Study data with the Baseline data at pre-randomization of the Core Study.
Time Frame: Baseline; up to Week 260
Population: ITT Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 2 | 2
Score on a scale | 0.00 (0.00) | 0.00 (0.00)

38. Secondary Outcome: Mean Change From the Pre-randomization Baseline of the Core Study to the End of Treatment in D-KEFS Number-letter Switching Completion Time Scaled Score
Description: D-KEFS Number-letter Switching Completion Time Scale was used to measure cognitive flexibility, task-set switching, and general executive functioning. The raw score i.e., total time in seconds for completing the number-letter switching trial was measured in the range of 0-240; higher scores indicated worse functioning. The raw score was normed with a referenced score to calculate a scaled score (i.e., score on a scale) ranging from 1-19; higher scores indicated better functioning. Change from the pre-randomization Baseline of the core study to the End of Treatment are reported as score on a scale. Negative values indicate worsening and positive values indicate improvement in cognitive function. The only data presented from the Core Studies in this report are the comparison of the Extension Study data with the Baseline data at pre-randomization of the Core Study.
Time Frame: Baseline; up to Week 260
Population: ITT Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 2 | 2
Score on a scale | 0.00 (0.00) | 0.00 (0.00)

39. Secondary Outcome: Mean Change From the Pre-randomization Baseline of the Core Study to the End of Treatment in D-KEFS Motor Speed Completion Time Scaled Score
Description: D-KEFS Motor Speed Completion Time Scale was used to measure motor speed. The raw score i.e., total time in seconds for completing the motor speed trial was measured in the range of 0-150; higher scores indicated worse functioning. The raw score was normed with a referenced score to calculate a scaled score (i.e., score on a scale) ranging from 1-19; higher scores indicated better motor speed. Change from the pre-randomization Baseline of the core study to the End of Treatment are reported as score on a scale. Negative values indicate worsening and positive values indicate improvement in motor speed. The only data presented from the Core Studies in this report are the comparison of the Extension Study data with the Baseline data at pre-randomization of the Core Study.
Time Frame: Baseline; up to Week 260
Population: ITT Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 2 | 3
Score on a scale | 0.00 (0.00) | -1.33 (2.309)

40. Secondary Outcome: Mean Change From the Pre-randomization Baseline of the Core Study to the End of Treatment in Purdue Pegboard Fine Motor Speed (Both Hands Z Score)
Description: Purdue Pegboard test was used to measure fine motor dexterity of both hands. The raw score was calculated as the total number of pegs in 30 seconds; higher scores indicated higher level of motor dexterity. The raw score was converted to a Z-score ranging from 0-19; higher scores indicate a higher level of motor dexterity. Change from the pre-randomization Baseline of the core study to the End of Treatment are reported as Z-score (i.e., score on a scale). Negative values indicate worsening and positive values indicate improvement in motor dexterity. The only data presented from the Core Studies in this report are the comparison of the Extension Study data with the Baseline data at pre-randomization of the Core Study.
Time Frame: Baseline; up to Week 260
Population: ITT Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Z Score
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 17 | 11
Z Score | 1.26 (3.272) | 9.55 (21.070)

41. Secondary Outcome: Mean Change From the Pre-randomization Baseline of the Core Study to the End of Treatment in Purdue Pegboard Fine Motor Speed (Dominant Hand Z Score)
Description: Purdue Pegboard test was used to measure fine motor dexterity of the dominant hand. The raw score was calculated as the total number of pegs in 30 seconds; higher scores indicated higher level of motor dexterity. The raw score was converted to a Z-score ranging from 0-19; higher scores indicate a higher level of motor dexterity. Change from the pre-randomization Baseline of the core study to the End of Treatment are reported as Z-score (i.e., score on a scale). Negative values indicate worsening and positive values indicate improvement in motor dexterity. The only data presented from the Core Studies in this report are the comparison of the Extension Study data with the Baseline data at pre-randomization of the Core Study.
Time Frame: Baseline; up to Week 260
Population: ITT Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Z Score
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 17 | 12
Z Score | 1.16 (3.192) | 9.23 (18.083)

42. Secondary Outcome: Mean Change From the Pre-randomization Baseline of the Core Study to the End of Treatment in Purdue Pegboard Fine Motor Speed (Non Dominant Hand Z Score)
Description: Purdue Pegboard test was used to measure fine motor dexterity of the non dominant hand. The raw score was calculated as the total number of pegs in 30 seconds; higher scores indicated higher level of motor dexterity. The raw score was converted to a Z-score ranging from 0-19; higher scores indicate a higher level of motor dexterity. Change from the pre-randomization Baseline of the core study to the End of Treatment are reported as Z-score (i.e., score on a scale). Negative values indicate worsening and positive values indicate improvement in motor dexterity. The only data presented from the Core Studies in this report are the comparison of the Extension Study data with the Baseline data at pre-randomization of the Core Study.
Time Frame: Baseline; up to Week 260
Population: ITT Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Z Score
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 17 | 12
Z Score | 1.31 (3.329) | 10.21 (21.852)

43. Secondary Outcome: Mean Change From the Pre-randomization Baseline of the Core Study to the End of Treatment in Wechsler Adult Intelligence Scale (WAIS) Coding Scaled Score
Description: WAIS Coding Scale was used to measure processing speed. The raw score i.e., sum of correct substitutions was measured in the range of 0-16. The raw score was normed with a referenced score to calculate a scaled score (i.e., score on a scale) ranging from 1-19; higher scores indicated better processing speed. Change from the pre-randomization Baseline of the core study to the End of Treatment are reported as score on a scale. Negative values indicate worsening and positive values indicate improvement in processing speed. The only data presented from the Core Studies in this report are the comparison of the Extension Study data with the Baseline data at pre-randomization of the Core Study.
Time Frame: Baseline; up to Week 260
Population: ITT Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 0 | 2
Score on a scale |  | 0.00 (0.00)

44. Secondary Outcome: Mean Change From the Pre-randomization Baseline of the Core Study to the End of Treatment in WAIS Digit Span Backward Scaled Score
Description: WAIS Digit Span Backward Scale was used to measure working memory. The raw score i.e., sum of correct trials was measured in the range of 0-16. The raw score was normed with a referenced score to calculate a scaled score (i.e., score on a scale) ranging from 1-19; higher scores indicated better working memory. Change from the pre-randomization Baseline of the core study to the End of Treatment are reported as score on a scale. Negative values indicate worsening and positive values indicate improvement in working memory. The only data presented from the Core Studies in this report are the comparison of the Extension Study data with the Baseline data at pre-randomization of the Core Study.
Time Frame: Baseline; up to Week 260
Population: ITT Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 315 | 366
Score on a scale
  Baseline: number analyzed (Participants) | 1 | 8
  Baseline | 0.0 (NA) — Standard deviation was not calculated for a single participant. | 0.0 (0.0)
  Week 48: number analyzed (Participants) | 1 | 4
  Week 48 | 0.0 (NA) — Standard deviation was not calculated for a single participant. | 0.25 (0.50)
  End of Treatment: number analyzed (Participants) | 0 | 7
  End of Treatment |  | -0.14 (0.378)

45. Secondary Outcome: Mean Change From the Pre-randomization Baseline of the Core Study to the End of Treatment in WAIS Digit Span Forward Scaled Score
Description: WAIS Digit Span Forward Scale was used to measure auditory memory. The raw score i.e., sum of correct trials was measured in the range of 0-16. The raw score was normed with a referenced score to calculate a scaled score (i.e., score on a scale) ranging from 1-19; higher scores indicated better auditory memory. Change from the pre-randomization Baseline of the core study to the End of Treatment are reported as score on a scale. Negative values indicate worsening and positive values indicate improvement in auditory memory. The only data presented from the Core Studies in this report are the comparison of the Extension Study data with the Baseline data at pre-randomization of the Core Study.
Time Frame: Baseline; up to Week 260
Population: ITT Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 315 | 366
Score on a scale
  Baseline: number analyzed (Participants) | 1 | 8
  Baseline | 0.0 (NA) — Standard deviation was not calculated for a single participant. | 0.13 (1.808)
  Week 48: number analyzed (Participants) | 1 | 4
  Week 48 | 0.0 (NA) — Standard deviation was not calculated for a single participant. | -0.25 (1.258)
  End of Treatment: number analyzed (Participants) | 0 | 7
  End of Treatment |  | 0.14 (2.268)

46. Secondary Outcome: Mean Change From the Pre-randomization Baseline of the Core Study to the End of Treatment in WAIS Longest Digit Span Backward Scaled Score
Description: WAIS Longest Digit Span Backward Scale was used to measure working memory. The raw score i.e., sum of correct trials was measured in the range of 2-8. The raw score was normed with a referenced score to calculate a scaled score (i.e., score on a scale) ranging from 1-19; higher scores indicated better working memory. Change from the pre-randomization Baseline of the core study to the End of Treatment are reported as score on a scale. Negative values indicate worsening and positive values indicate improvement in working memory. The only data presented from the Core Studies in this report are the comparison of the Extension Study data with the Baseline data at pre-randomization of the Core Study.
Time Frame: Baseline; up to Week 260
Population: ITT Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 315 | 366
Score on a scale
  Baseline: number analyzed (Participants) | 1 | 8
  Baseline | 0.00 (NA) — Standard deviation was not calculated for a single participant. | 0.00 (0.00)
  Week 48: number analyzed (Participants) | 1 | 4
  Week 48 | 0.00 (NA) — Standard deviation was not calculated for a single participant. | 0.00 (0.00)
  End of Treatment: number analyzed (Participants) | 0 | 7
  End of Treatment |  | 0.00 (0.00)

47. Secondary Outcome: Mean Change From the Pre-randomization Baseline of the Core Study to the End of Treatment in WAIS Longest Digit Span Forward Scaled Score
Description: WAIS Longest Digit Span Forward Scale was used to measure auditory memory. The raw score i.e., sum of correct trials was measured in the range of 2-8. The raw score was normed with a referenced score to calculate a scaled score (i.e., score on a scale) ranging from 1-19; higher scores indicated better auditory memory. Change from the pre-randomization Baseline of the core study to the End of Treatment are reported as score on a scale. Negative values indicate worsening and positive values indicate improvement in auditory memory. The only data presented from the Core Studies in this report are the comparison of the Extension Study data with the Baseline data at pre-randomization of the Core Study.
Time Frame: Baseline; up to Week 260
Population: ITT Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 315 | 366
Score on a scale
  Baseline: number analyzed (Participants) | 1 | 8
  Baseline | 0.0 (NA) — Standard deviation was not calculated for a single participant. | 0.13 (1.642)
  Week 48: number analyzed (Participants) | 1 | 4
  Week 48 | 0.0 (NA) — Standard deviation was not calculated for a single participant. | 0.25 (1.258)
  End of Treatment: number analyzed (Participants) | 0 | 7
  End of Treatment |  | -0.14 (1.574)

48. Secondary Outcome: Mean Change From the Pre-randomization Baseline of the Core Study to the End of Treatment in Wechsler Abbreviated Scale of Intelligence (WASI)-II Vocabulary T Score
Description: WAIS-II Vocabulary T Score was used to estimate general intellectual ability based on fund of information and verbal intelligence. The raw score i.e., the sum of correct responses was converted to a T-score ranging from 20-80 using the WASI assessment manual; T-scores are standard scores with a mean of 50 and a standard deviation of 10. Higher scores indicate a higher level of intelligence. Change from the pre-randomization Baseline of the core study to the End of Treatment are reported as T-score (i.e., score on a scale). Negative values indicate worsening and positive values indicate improvement in intelligence. The only data presented from the Core Studies in this report are the comparison of the Extension Study data with the Baseline data at pre-randomization of the Core Study.
Time Frame: Baseline; up to Week 260
Population: ITT Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: T Score
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 4 | 6
T Score | 0.00 (0.00) | -4.00 (12.247)

49. Secondary Outcome: Mean Change From the Pre-randomization Baseline of the Core Study to the End of Treatment in WASI-II Matrix Reasoning T Score
Description: WASI-II Matrix Reasoning T Score was used to estimate general intellectual ability based abstract reasoning. The raw score i.e., the sum of correct responses was converted to a T-score ranging from 20-80 using the WASI assessment manual; T-scores are standard scores with a mean of 50 and a standard deviation of 10. Higher scores indicate a higher level of abstract reasoning. Change from the pre-randomization Baseline of the core study to the End of Treatment are reported as T-score (i.e., score on a scale). Negative values indicate worsening and positive values indicate improvement in abstract reasoning. The only data presented from the Core Studies in this report are the comparison of the Extension Study data with the Baseline data at pre-randomization of the Core Study.
Time Frame: Baseline; up to Week 260
Population: ITT Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: T Score
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 4 | 7
T Score | -1.50 (3.000) | -3.29 (5.376)

50. Secondary Outcome: Mean Change From the Pre-randomization Baseline of the Core Study to the End of Treatment in Wechsler Intelligence Scale for Children (WISC) Coding Scaled Score
Description: WISC Coding Scale was used to measure processing speed in children aged 6-16 years 11 months, with scores ranging from 0 to 119. Higher scores indicate better processing speed. Change from the pre-randomization Baseline of the core study to the End of Treatment are reported as score on a scale. Negative values indicate worsening and positive values indicate improvement in processing speed. The only data presented from the Core Studies in this report are the comparison of the Extension Study data with the Baseline data at pre-randomization of the Core Study.
Time Frame: Baseline; up to Week 260
Population: ITT Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 5 | 0
Score on a scale | -0.40 (1.817) |

51. Secondary Outcome: Mean Change From the Pre-randomization Baseline of the Core Study to the End of Treatment in WISC Digit Span Backward Scaled Score
Description: WISC Digit Span Backward Scale was used to measure working memory. The raw score i.e., sum of correct trials was measured on a scale of 0-18; higher scores indicated better working memory. Change from the pre-randomization Baseline of the core study to the End of Treatment are reported as score on a scale. Negative values indicate worsening and positive values indicate improvement in working memory. The only data presented from the Core Studies in this report are the comparison of the Extension Study data with the Baseline data at pre-randomization of the Core Study.
Time Frame: Baseline; up to Week 260
Population: ITT Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 6 | 0
Score on a scale | 0.00 (0.632) |

52. Secondary Outcome: Mean Change From the Pre-randomization Baseline of the Core Study to the End of Treatment in WISC Digit Span Forward Scaled Score
Description: WISC Digit Span Forward Scale was used to measure auditory memory. The raw score i.e., sum of correct trials was measured on a scale of 0-18; higher scores indicated better auditory memory. Change from the pre-randomization Baseline of the core study to the End of Treatment are reported as score on a scale. Negative values indicate worsening and positive values indicate improvement in auditory memory. The only data presented from the Core Studies in this report are the comparison of the Extension Study data with the Baseline data at pre-randomization of the Core Study.
Time Frame: Baseline; up to Week 260
Population: ITT Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 7 | 0
Score on a scale | 0.57 (0.787) |

53. Secondary Outcome: Mean Change From the Pre-randomization Baseline of the Core Study to the End of Treatment in WISC Longest Digit Span Backward Scaled Score
Description: WISC Longest Digit Span Backward Scale was used to measure working memory. The raw score i.e., sum of correct trials was measured on a scale of 2-8; higher scores indicated better working memory. Change from the pre-randomization Baseline of the core study to the End of Treatment are reported as score on a scale. Negative values indicate worsening and positive values indicate improvement in working memory. The only data presented from the Core Studies in this report are the comparison of the Extension Study data with the Baseline data at pre-randomization of the Core Study.
Time Frame: Baseline; up to Week 260
Population: ITT Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 6 | 0
Score on a scale | 0.00 (1.265) |

54. Secondary Outcome: Mean Change From the Pre-randomization Baseline of the Core Study to the End of Treatment in WISC Longest Digit Span Forward Scaled Score
Description: WISC Longest Digit Span Forward Scale was used to measure auditory memory. The raw score i.e., sum of correct trials was measured on a scale of 2-10; higher scores indicated better auditory memory. Change from the pre-randomization Baseline of the core study to the End of Treatment are reported as score on a scale. Negative values indicate worsening and positive values indicate improvement in auditory memory. The only data presented from the Core Studies in this report are the comparison of the Extension Study data with the Baseline data at pre-randomization of the Core Study.
Time Frame: Baseline; up to Week 260
Population: ITT Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 6 | 0
Score on a scale | 0.17 (0.408) |

55. Secondary Outcome: Mean Change From the Pre-randomization Baseline of the Core Study to the End of Treatment in Wechsler Preschool & Primary Scale of Intelligence (WPPSI)-IV Bug Search T Score
Description: WPPSI-IV Bug Search T Score was used to measure processing speed and complex attention. The raw score i.e., the sum of correct responses was measured on a scale of 1-19 and converted to a T-score ranging from 20-80; T-scores are standard scores with a mean of 50 and a standard deviation of 10. Higher scores indicate a higher level of attention. Change from the pre-randomization Baseline of the core study to the End of Treatment are reported as T-score (i.e., score on a scale). Negative values indicate worsening and positive values indicate improvement in attention. The only data presented from the Core Studies in this report are the comparison of the Extension Study data with the Baseline data at pre-randomization of the Core Study.
Time Frame: Baseline; up to Week 260
Population: ITT Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: T Score
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 315 | 0
T Score
  Baseline: number analyzed (Participants) | 2 | 0
  Baseline | 0.0 (0.0) |
  Week 48: number analyzed (Participants) | 1 | 0
  Week 48 | 0.0 (NA) — Standard deviation was not calculated for a single participant. |
  End of Treatment: number analyzed (Participants) | 0 | 0

56. Secondary Outcome: Mean Change From the Pre-randomization Baseline of the Core Study to the End of Treatment in WPPSI-IV Receptive Vocabulary T Score
Description: WPPSI-IV Receptive Vocabulary T Score was used to measure fund of information. The raw score i.e., the sum of correct responses was measured on a scale of 1-19 and converted to a T-score ranging from 20-80; T-scores are standard scores with a mean of 50 and a standard deviation of 10. Higher scores indicate a higher level of intelligence. Change from the pre-randomization Baseline of the core study to the End of Treatment are reported as as T-score (i.e., score on a scale). Negative values indicate worsening and positive values indicate improvement in intelligence. The only data presented from the Core Studies in this report are the comparison of the Extension Study data with the Baseline data at pre-randomization of the Core Study.
Time Frame: Baseline; up to Week 260
Population: ITT Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: T Score
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 0 | 1
T Score |  | -1.00 (NA) — Standard deviation was not calculated for a single participant.

57. Secondary Outcome: Mean Change From the Pre-randomization Baseline of the Core Study to the End of Treatment in WPPSI-IV Matrix Reasoning T Score
Description: WPPSI-IV Matrix Reasoning T Score was used to measure abstract reasoning. The raw score i.e., the sum of correct responses was measured on a scale of 1-19 and converted to a T-score ranging from 20-80; T-scores are standard scores with a mean of 50 and a standard deviation of 10. Higher scores indicate a higher level of abstract reasoning. Change from the pre-randomization Baseline of the core study to the End of Treatment are reported as T-score (i.e., score on a scale). Negative values indicate worsening and positive values indicate improvement in abstract reasoning. The only data presented from the Core Studies in this report are the comparison of the Extension Study data with the Baseline data at pre-randomization of the Core Study.
Time Frame: Baseline; up to Week 260
Population: ITT Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: T Score
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 315 | 366
T Score
  Baseline: number analyzed (Participants) | 4 | 1
  Baseline | 0.75 (6.994) | -19.0 (NA) — Standard deviation was not calculated for a single participant.
  Week 48: number analyzed (Participants) | 4 | 0
  Week 48 | -0.75 (6.994) |
  End of Treatment: number analyzed (Participants) | 0 | 0

58. Secondary Outcome: Mean Change From the Pre-randomization Baseline of the Core Study to the End of Treatment in Expressive One-Word Picture Vocabulary Test (EOWPVT) Scaled Score
Description: Expressive One-Word Picture Vocabulary Test-4th edition was used to test vocabulary. The raw score i.e., the sum of correct responses was measured on a scale of 1-19 and converted to a T-score ranging from 0-83; T-scores are standard scores with a mean of 100 and a standard deviation of 15. Higher scores indicate a higher level of language performance. Change from the pre-randomization Baseline of the core study to the End of Treatment are reported as as T-score (i.e., score on a scale). Negative values indicate worsening and positive values indicate improvement in language performance. The only data presented from the Core Studies in this report are the comparison of the Extension Study data with the Baseline data at pre-randomization of the Core Study.
Time Frame: Baseline; up to Week 260
Population: ITT Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 2 | 2
T score | -31.00 (56.569) | -31.00 (53.740)

59. Secondary Outcome: Mean Change From the Pre-randomization Baseline of the Core Study to the End of Treatment in a Developmental NEuroPSYchological Assessment (NEPSY)-2 Word Generation Scaled Score
Description: Developmental NEuroPSYchological Assessment (NEPSY)-2 Word Generation Scale was used to measure verbal fluency. The raw score i.e., the sum of correct responses was converted to a scaled score (i.e., score on a scale) ranging from 1-19; higher scores indicate a higher level of verbal fluency. Change from the pre-randomization Baseline of the core study to the End of Treatment are reported as score on a scale. Negative values indicate worsening and positive values indicate improvement in verbal fluency. The only data presented from the Core Studies in this report are the comparison of the Extension Study data with the Baseline data at pre-randomization of the Core Study.
Time Frame: Baseline; up to Week 260
Population: ITT Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 2 | 1
Score on a scale | -1.00 (1.414) | 3.39 (NA) — Standard deviation was not calculated for a single participant.

60. Secondary Outcome: Mean Change From the Pre-randomization Baseline of the Core Study to the End of Treatment in Visual Perception Standard Scaled Score
Description: Visual Perception Standard scale was used to measure visual motor functioning. The raw score i.e., the sum of the correct responses was measured on a 6-standard score range. Score range of 70-79 indicated "low," 80-89 indicated "below average," 90-109 indicated "average," 110-119 indicated "above average," 120-129 indicated "high," and >129 indicated "very high" visual motor functioning. Change from the pre-randomization Baseline of the core study to the End of Treatment are reported as score on a scale. Negative values indicate worsening and positive values indicate improvement in visual motor functioning. The only data presented from the Core Studies in this report are the comparison of the Extension Study data with the Baseline data at pre-randomization of the Core Study.
Time Frame: Baseline; up to Week 260
Population: ITT Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
Number analyzed (Participants) | 1 | 3
Score on a scale | 0.00 (NA) — Standard deviation was not calculated for a single participant. | 2.67 (7.767)

ADVERSE EVENTS:
Time Frame: Up to Week 260
Description: Treatment-emergent adverse events (TEAEs), defined as adverse events (AEs) that started, worsened in severity or seriousness, following the first dose of investigational medicinal product in this study, whether or not considered related to the participant's participation in the research, are reported. Any AEs that continued from the Core Study were only classified as treatment emergent if they worsened in this study.
Arm/Group | Dravet Syndrome | Lennox-Gastaut Syndrome
All-Cause Mortality (participants affected / at risk) | 6/315 | 12/366
Serious Adverse Events (participants affected / at risk) | 133/315 | 157/366
Other Adverse Events (participants affected / at risk) | 292/315 | 338/366
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dravet Syndrome (N=315) | Lennox-Gastaut Syndrome (N=366)
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 | 1
Eosinophilia (Blood and lymphatic system disorders) | 0 | 1
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 3 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Rett's disorder (Congenital, familial and genetic disorders) | 0 | 1
Blindness transient (Eye disorders) | 0 | 1
Eye oedema (Eye disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 5 | 5
Faecaloma (Gastrointestinal disorders) | 1 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 2
Haematochezia (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 4
Ileus paralytic (Gastrointestinal disorders) | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 3
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 3
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2
Tooth loss (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 13
Asthenia (General disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Device dislocation (General disorders) | 0 | 1
Device malfunction (General disorders) | 0 | 1
Drowning (General disorders) | 1 | 0
Drug withdrawal syndrome (General disorders) | 0 | 1
Effusion (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Generalised oedema (General disorders) | 0 | 1
Hypothermia (General disorders) | 0 | 2
Malaise (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 17 | 11
Sudden unexplained death in epilepsy (General disorders) | 4 | 4
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 0
Hepatitis acute (Hepatobiliary disorders) | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0
Abdominal wall abscess (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 2 | 1
Appendicitis perforated (Infections and infestations) | 1 | 0
Atypical pneumonia (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 2
Bronchitis (Infections and infestations) | 1 | 0
Campylobacter gastroenteritis (Infections and infestations) | 0 | 1
Catheter site abscess (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 2
Cellulitis staphylococcal (Infections and infestations) | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1
Colon gangrene (Infections and infestations) | 0 | 1
Corona virus infection (Infections and infestations) | 1 | 0
Croup infectious (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 0 | 1
Empyema (Infections and infestations) | 0 | 1
Enterococcal infection (Infections and infestations) | 1 | 0
Enterovirus infection (Infections and infestations) | 2 | 0
Epstein-Barr virus infection (Infections and infestations) | 1 | 0
Escherichia infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 4 | 2
Infected bites (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Infectious mononucleosis (Infections and infestations) | 1 | 0
Infective myositis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 7 | 3
Klebsiella infection (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 5
Lower respiratory tract infection (Infections and infestations) | 2 | 1
Meningitis viral (Infections and infestations) | 1 | 0
Metapneumovirus infection (Infections and infestations) | 1 | 1
Myelitis (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1
Otitis externa (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 0 | 2
Otitis media acute (Infections and infestations) | 0 | 1
Parainfluenzae virus infection (Infections and infestations) | 2 | 2
Peritonitis (Infections and infestations) | 0 | 1
Pertussis (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 2 | 1
Pneumonia (Infections and infestations) | 20 | 26
Pneumonia bacterial (Infections and infestations) | 1 | 1
Pneumonia influenzal (Infections and infestations) | 0 | 1
Pneumonia pseudomonal (Infections and infestations) | 0 | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 | 0
Pneumonia staphylococcal (Infections and infestations) | 1 | 1
Pneumonia viral (Infections and infestations) | 2 | 2
Pseudomonas infection (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 1
Rectal abscess (Infections and infestations) | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 4 | 0
Respiratory tract infection (Infections and infestations) | 1 | 2
Respiratory tract infection viral (Infections and infestations) | 1 | 0
Rhinovirus infection (Infections and infestations) | 3 | 2
Sepsis (Infections and infestations) | 0 | 6
Septic shock (Infections and infestations) | 1 | 2
Sinusitis (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 2
Superinfection (Infections and infestations) | 0 | 1
Superinfection bacterial (Infections and infestations) | 1 | 0
Tracheitis (Infections and infestations) | 0 | 1
Tracheobronchitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 2
Urinary tract infection (Infections and infestations) | 1 | 9
Viral infection (Infections and infestations) | 1 | 3
Viral pharyngitis (Infections and infestations) | 1 | 1
Viral upper respiratory tract infection (Infections and infestations) | 3 | 1
West Nile viral infection (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Ear injury (Injury, poisoning and procedural complications) | 0 | 1
Extradural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Eye contusion (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 3
Feeding tube complication (Injury, poisoning and procedural complications) | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0
Near drowning (Injury, poisoning and procedural complications) | 2 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Skull fracture (Injury, poisoning and procedural complications) | 1 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Tooth avulsion (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 2
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 7 | 7
Ammonia increased (Investigations) | 1 | 0
Anticonvulsant drug level increased (Investigations) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 10 | 6
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0
Body temperature fluctuation (Investigations) | 0 | 1
Eosinophil count increased (Investigations) | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 4 | 3
Gastrointestinal stoma output increased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 2 | 6
International normalised ratio increased (Investigations) | 1 | 0
Lipase increased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 1 | 2
Norovirus test positive (Investigations) | 1 | 0
Oxygen consumption increased (Investigations) | 0 | 1
Oxygen saturation decreased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 1 | 0
Transaminases abnormal (Investigations) | 0 | 1
Transaminases increased (Investigations) | 2 | 5
Weight decreased (Investigations) | 1 | 4
Decreased appetite (Metabolism and nutrition disorders) | 0 | 3
Dehydration (Metabolism and nutrition disorders) | 6 | 5
Enteral feeding intolerance (Metabolism and nutrition disorders) | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2
Hypophagia (Metabolism and nutrition disorders) | 0 | 2
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 3
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 | 1
Metabolic disorder (Metabolism and nutrition disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Altered state of consciousness (Nervous system disorders) | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 1
Cerebral atrophy (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 34 | 44
Depressed level of consciousness (Nervous system disorders) | 0 | 2
Dyskinesia (Nervous system disorders) | 1 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 2 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 4 | 1
Hemiparesis (Nervous system disorders) | 0 | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 3 | 2
Metabolic encephalopathy (Nervous system disorders) | 0 | 1
Movement disorder (Nervous system disorders) | 0 | 1
Myoclonic epilepsy (Nervous system disorders) | 0 | 1
Myoclonus (Nervous system disorders) | 1 | 0
Neuromyopathy (Nervous system disorders) | 0 | 1
Partial seizures (Nervous system disorders) | 1 | 0
Postictal state (Nervous system disorders) | 1 | 0
Sedation (Nervous system disorders) | 0 | 1
Seizure cluster (Nervous system disorders) | 2 | 1
Somnolence (Nervous system disorders) | 2 | 1
Status epilepticus (Nervous system disorders) | 47 | 42
Abnormal behaviour (Psychiatric disorders) | 2 | 1
Aggression (Psychiatric disorders) | 1 | 2
Agitation (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1
Hallucinations, mixed (Psychiatric disorders) | 1 | 0
Irritability (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 6
Self injurious behaviour (Psychiatric disorders) | 0 | 1
Sleep disorder (Psychiatric disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Nephrocalcinosis (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal cyst (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 5
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 3
Testicular torsion (Reproductive system and breast disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 10
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Choking (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 9
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 4 | 16
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 6
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 8
Respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 0 | 1
Child abuse (Social circumstances) | 0 | 1
Foot operation (Surgical and medical procedures) | 0 | 1
Gastrostomy (Surgical and medical procedures) | 0 | 1
Hypotension (Vascular disorders) | 0 | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dravet Syndrome (N=315) | Lennox-Gastaut Syndrome (N=366)
Constipation (Gastrointestinal disorders) | 20 | 41
Diarrhoea (Gastrointestinal disorders) | 133 | 138
Nausea (Gastrointestinal disorders) | 16 | 30
Vomiting (Gastrointestinal disorders) | 63 | 99
Fatigue (General disorders) | 38 | 38
Bronchitis (Infections and infestations) | 14 | 23
Pyrexia (General disorders) | 117 | 123
Ear infection (Infections and infestations) | 35 | 50
Gastroenteritis (Infections and infestations) | 16 | 6
Gastroenteritis viral (Infections and infestations) | 11 | 29
Influenza (Infections and infestations) | 31 | 42
Nasopharyngitis (Infections and infestations) | 78 | 58
Otitis media (Infections and infestations) | 21 | 21
Pharyngitis streptococcal (Infections and infestations) | 24 | 26
Sinusitis (Infections and infestations) | 38 | 48
Pneumonia (Infections and infestations) | 22 | 31
Upper respiratory tract infection (Infections and infestations) | 77 | 102
Urinary tract infection (Infections and infestations) | 18 | 47
Viral upper respiratory tract infection (Infections and infestations) | 9 | 19
Contusion (Injury, poisoning and procedural complications) | 15 | 24
Fall (Injury, poisoning and procedural complications) | 20 | 20
Laceration (Injury, poisoning and procedural complications) | 8 | 35
Alanine aminotransferase increased (Investigations) | 31 | 23
Aspartate aminotransferase increased (Investigations) | 30 | 13
Gamma-glutamyltransferase increased (Investigations) | 29 | 18
Weight decreased (Investigations) | 20 | 58
Decreased appetite (Metabolism and nutrition disorders) | 99 | 92
Convulsion (Nervous system disorders) | 60 | 120
Drooling (Nervous system disorders) | 11 | 21
Headache (Nervous system disorders) | 18 | 26
Lethargy (Nervous system disorders) | 19 | 32
Sedation (Nervous system disorders) | 16 | 27
Somnolence (Nervous system disorders) | 86 | 106
Abnormal behaviour (Psychiatric disorders) | 32 | 22
Aggression (Psychiatric disorders) | 19 | 29
Insomnia (Psychiatric disorders) | 16 | 40
Irritability (Psychiatric disorders) | 26 | 28
Cough (Respiratory, thoracic and mediastinal disorders) | 42 | 63
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 13 | 46
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 19 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-04-25): https://cdn.clinicaltrials.gov/large-docs/73/NCT02224573/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-06): https://cdn.clinicaltrials.gov/large-docs/73/NCT02224573/SAP_001.pdf